CLINICAL TRIAL: NCT02321384
Title: A Single-Center, Randomized, Double-Blind, Single and Multiple Ascending Dose, Placebo-Controlled Study to Investigate the Safety, Tolerability and Pharmacokinetics of RO6889678 and the Combination of RO6889678 With Ritonavir Following Oral Administration, the Effect of Food on the Pharmacokinetics of RO6889678 and the Effect of Multiple Oral Dosing of RO6889678 and the Combination of RO6889678 With Ritonavir on the Pharmacokinetics of Midazolam in Healthy Subjects
Brief Title: A Study to Investigate the Safety, Tolerability and Pharmacokinetics of RO6889678 and the Combination of RO6889678 With Ritonavir in Healthy Participants
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: NP29454; 2014-002297-36 (EudraCT Number)
Record Dates: First submitted 2014-12-17; First posted 2014-12-22 (Estimated); Last update posted 2017-04-05 (Actual); Status verified 2017-04

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — Midazolam; Ritonavir

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- A: SAD Cohorts - RO6889678/Matching Placebo (Experimental): Healthy participants will be enrolled into 1 of 6 planned SAD cohorts to receive single dose of RO6889678/matching placebo in fasted state as per anticipated dose escalation sequence (30 milligrams [mg], 100 mg, 300 mg, 600 mg, 1000 mg and 1500 mg). Cohort 1 will be split in 2 groups: 2 participants will be dosed 1 day (1 on RO6889678 and 1 on matching placebo) and 3 participants (2 on RO6889678 and 1 on matching placebo) will be dosed at least 24 hours afterward following satisfactory safety assessment for first 2 participants. Cohort 2 & beyond will include 8 healthy participants with 6 participants randomly assigned to RO6889678 & 2 randomly assigned to placebo. Participants who will tolerate fasted dose and agree to continue in food-effect SAD cohort, will receive single dose (dose level, either 300 mg or 600 mg, decided based on PK and safety data of first 2 SAD cohorts) of RO6889678/matching placebo with US FDA recommended high-fat and high-calorie breakfast on Day 16.
  Interventions: Drug: Placebo; Drug: RO6889678
- B: MAD Cohorts - RO6889678/Matching Placebo (Experimental): Healthy participants will be enrolled into 1 of 4 planned MAD cohorts to receive RO6889678 or matching placebo (at a dose that will be decided as per the safety, tolerability and PK data from SAD 4 cohort) twice daily (BID) for 14 days except for Day 14, where only one dose in the morning will be given. Each of the MAD cohorts will include 8 healthy participants with 6 participants randomly assigned to RO6889678 and 2 participants randomly assigned to placebo. All participants enrolled to the MAD cohorts will receive an oral microdose of midazolam (100 micrograms [mcg]) before (Day -1) and after (Day 14) the repeat treatment with RO6889678 or matching placebo.
  Interventions: Drug: Placebo; Drug: RO6889678; Drug: Midazolam
- C:RTV-Boosted SAD & MAD Cohorts-RO6889678/Matching Placebo+RTV (Experimental): Healthy participants will be enrolled in up to 3 SAD cohorts (2 compulsory and 1 optional) and up to 3 MAD cohorts (1 compulsory and 2 optional) to receive RO6889678 in combination with RTV in fed state. Participants of the first 2 RTV-boosted SAD cohorts will receive 100 mg RO6889678 + 100 mg RTV and 300 mg RO6889678 + 100 mg RTV respectively. Based on the PK and safety evaluation of the first 2 RTV-boosted SAD cohorts, another SAD cohort may be enrolled to receive a different dose of RO6889678 in combination with RTV. MAD RTV-boosted cohort will start based on the safety, tolerability and PK data of the RTV-boosted SAD cohorts. All participants enrolled to the RTV-boosted MAD cohorts will receive RO6889678 or placebo together with RTV on BID schedule for 14 days, and additionally an oral microdose of midazolam (100 mcg) before (Day -1) and after (Day 14) the treatment.
  Interventions: Drug: Placebo; Drug: RO6889678; Drug: Midazolam; Drug: Ritonavir

INTERVENTIONS:
Drug: Placebo — Placebo matched to RO6889678 will be administered orally as a single dose on Day 1 in SAD cohorts and multiple doses BID from Day 1 to Day 14 (no second BID dose on Day 14) in MAD cohorts.
Drug: RO6889678 — RO6889678 will be administered orally as a single dose on Day 1 in SAD cohorts and multiple doses BID from Day 1 to Day 14 (no second BID dose on Day 14) in MAD cohorts.
Drug: Midazolam — Single dose of 100 mcg midazolam solution will be administered orally, before (Day -1) and after (Day 14) the treatment with RO6889678 or matching placebo.
  Arms: B: MAD Cohorts - RO6889678/Matching Placebo; C:RTV-Boosted SAD & MAD Cohorts-RO6889678/Matching Placebo+RTV
Drug: Ritonavir — RTV will be administered orally as a single dose on Day 1 in RTV-boosted SAD cohorts and multiple doses BID from Day 1 to Day 14 (no second BID dose on Day 14) in RTV-boosted MAD cohorts.
  Arms: C:RTV-Boosted SAD & MAD Cohorts-RO6889678/Matching Placebo+RTV

SUMMARY:
This study is a single-center, double-blind, randomized, placebo-controlled, single-ascending dose (SAD) and multiple-ascending dose (MAD) study that will evaluate the safety, tolerability and pharmacokinetics (PK) of RO6889678 and the combination of RO6889678 with Ritonavir (RTV) following oral administration in healthy volunteers. The effect of food on the PK of RO6889678 and the effect of multiple dosing of RO6889678 and the combination of RO6889678 with RTV on the PK of a single oral microdose of midazolam will be evaluated.

Healthy participants will be screened up to 28 days before randomization and sequentially enrolled into SAD and MAD unboosted and RTV-boosted cohorts, then randomly assigned to RO6889678 or matching placebo. In RTV-boosted cohorts participants will take RO6889678 in combination with RTV. To explore the effect of food on RO6889678 PK, a cohort of volunteers will participate in a two-period food effect sub-study. Participants enrolled in the MAD cohorts will be given an oral microdose of midazolam before and after the repeat treatment with RO6889678 to evaluate the drug-drug interaction potential of RO6889678.

ELIGIBILITY:
Inclusion Criteria:

* Absence of evidence of any active or chronic disease following a detailed medical and surgical history, a complete physical examination including vital signs, 12-lead Electrocardiogram (ECG), hematology, blood chemistry, serology and urinalysis
* A Body Mass Index (BMI) between 18 to 30 kilograms per square meter (kg/m^2), inclusive
* Female participants must be either surgically sterile (by means of hysterectomy and/or bilateral oophorectomy) or post-menopausal for at least one year (defined as amenorrhea greater than or equal to [>/=] 12 consecutive months without another cause, and confirmed by follicle stimulating hormone level greater than [>] 35 milli-international units per milliliter [mIU/mL])
* Male participants must agree to use two adequate methods of contraception with their female partners of childbearing potential, including a barrier method during the treatment period and for at least 2 months after the last dose of study drug

Exclusion Criteria:

* History or symptoms of any significant disease
* Pregnant or lactating
* Personal or family history of congenital long QT syndrome or sudden death
* Significant acute infection, e.g. influenza, local infection, acute gastrointestinal symptoms or any other clinically significant illness within two weeks of dose administration
* Clinically relevant ECG abnormalities on screening ECG
* Participation in an investigational drug or device study within 90 days prior to screening
* Medical or social conditions that would potentially interfere with the participant's ability to comply with the study visit schedule or the study assessments

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2014-12-15 (Actual); Primary Completion 2015-11-26 (Actual); Study Completion 2015-11-26 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Adverse Events | From screening to the end of follow-up (up to 12 weeks)
SAD Cohort: Maximum Observed Plasma Concentration (Cmax) of RO6889678 | Pre-dose (0 hour [hr]) on Day 1; 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72 and 96 hr post Day 1 dose
SAD Cohort: Time to Reach Cmax (Tmax) of RO6889678 | Pre-dose (0 hr) on Day 1; 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72 and 96 hr post Day 1 dose
Outcome Measure: SAD Cohort: Area Under the Plasma Concentration Versus Time Curve up to the Last Measurable Concentration (AUC0-last) of RO6889678 | Pre-dose (0 hr) on Day 1; 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72 and 96 hr post Day 1 dose
SAD Cohort: Area Under the Plasma Concentration Versus Time Curve Extrapolated to Infinity (AUC0-inf) of RO6889678 | Pre-dose (0 hr) on Day 1; 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72 and 96 hr post Day 1 dose
SAD Cohort: Apparent Terminal Half-life (t1/2) of RO6889678 | Pre-dose (0 hr) on Day 1; 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72 and 96 hr post Day 1 dose
SAD Cohort: Apparent Oral Clearance (CL/F) of RO6889678 | Pre-dose (0 hr) on Day 1; 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72 and 96 hr post Day 1 dose
RO6889678 Only SAD Cohort 3 and 6 and all RTV-Boosted SAD Cohorts: Cumulative Amount Excreted Unchanged in Urine (Ae) of RO6889678 | Pre-dose (0 hr) on Day 1; 0-4, 4-8, 8-12, 12-24, 24-48 hours post Day 1 dose
RO6889678 Only SAD Cohort 3 and 6 and all RTV-Boosted SAD Cohorts: Renal Clearance (CLR) of RO6889678 | Pre-dose (0 hr) on Day 1; 0-4, 4-8, 8-12, 12-24, 24-48 hours post Day 1 dose
MAD Cohort: Cmax of RO6889678 | Pre-dose (0 hr), 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10 & 12 hr after first dose on Day 1; pre-dose (0 hr before morning dose) on Days 2, 3, 4, 5, 7; and pre-dose (0 hr), 0.25,0.5,1,1.5,2,3,4,6,8,10,12,24,36,48,72 & 96 hr after last morning dose on Day 14
MAD Cohort: Tmax of RO6889678 | Pre-dose (0 hr), 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10 & 12 hr after first dose on Day 1; pre-dose (0 hr before morning dose) on Days 2, 3, 4, 5, 7; and pre-dose (0 hr), 0.25,0.5,1,1.5,2,3,4,6,8,10,12,24,36,48,72 & 96 hr after last morning dose on Day 14
MAD Cohort: Area Under the Plasma Concentration Versus Time Curve for a Dosing Interval (AUC0-tau) of RO6889678 | Pre-dose (0 hr), 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10 & 12 hr after first dose on Day 1; pre-dose (0 hr before morning dose) on Days 2, 3, 4, 5, 7; and pre-dose (0 hr), 0.25,0.5,1,1.5,2,3,4,6,8,10,12,24,36,48,72 & 96 hr after last morning dose on Day 14
MAD Cohort: Plasma Trough Concentration (Ctrough) of RO6889678 | Pre-dose (0 hr before morning dose) on Days 2, 3, 4, 5, 7
MAD Cohort: Apparent Terminal Half-life (t1/2) of RO6889678 | Pre-dose (0 hr), 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10 & 12 hr after first dose on Day 1; pre-dose (0 hr before morning dose) on Days 2, 3, 4, 5, 7; and pre-dose (0 hr), 0.25,0.5,1,1.5,2,3,4,6,8,10,12,24,36,48,72 & 96 hr after last morning dose on Day 14
MAD Cohort: Accumulation Index of RO6889678 | Pre-dose (0 hr), 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10 & 12 hr after first dose on Day 1; pre-dose (0 hr before morning dose) on Days 2, 3, 4, 5, 7; and pre-dose (0 hr), 0.25,0.5,1,1.5,2,3,4,6,8,10,12,24,36,48,72 & 96 hr after last morning dose on Day 14
MAD Cohort: Ae of RO6889678 | Pre-dose (0 hr), 0-4, 4-8, 8-12 hours post morning dose on Day 1 and 14
MAD Cohort: CLR of RO6889678 | Pre-dose (0 hr), 0-4, 4-8, 8-12 hours post morning dose on Day 1 and 14
RTV-Boosted SAD Cohort: Cmax of RTV | Pre-dose (0 hr) on Day 1; 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72 and 96 hr post Day 1 dose
RTV-Boosted SAD Cohort: Tmax of RTV | Pre-dose (0 hr) on Day 1; 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72 and 96 hr post Day 1 dose
RTV-Boosted SAD Cohort: AUC0-last of RTV | Pre-dose (0 hr) on Day 1; 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72 and 96 hr post Day 1 dose
RTV-Boosted SAD Cohort: AUC0-inf of RTV | Pre-dose (0 hr) on Day 1; 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72 and 96 hr post Day 1 dose
RTV-Boosted SAD Cohort: Apparent Terminal t1/2 of RTV | Pre-dose (0 hr) on Day 1; 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72 and 96 hr post Day 1 dose
RTV-Boosted SAD Cohort: CL/F of RTV | Pre-dose (0 hr) on Day 1; 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72 and 96 hr post Day 1 dose
RTV-Boosted MAD Cohort: Cmax of RTV | Pre-dose (0 hr), 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10 & 12 hr after first dose on Day 1; pre-dose (0 hr before morning dose) on Days 2, 3, 4, 5, 7; and pre-dose (0 hr), 0.25,0.5,1,1.5,2,3,4,6,8,10,12,24,36,48,72 & 96 hr after last morning dose on Day 14
RTV-Boosted MAD Cohort: Tmax of RTV | Pre-dose (0 hr), 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10 & 12 hr after first dose on Day 1; pre-dose (0 hr before morning dose) on Days 2, 3, 4, 5, 7; and pre-dose (0 hr), 0.25,0.5,1,1.5,2,3,4,6,8,10,12,24,36,48,72 & 96 hr after last morning dose on Day 14
RTV-Boosted MAD Cohort: AUC0-tau of RTV | Pre-dose (0 hr), 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10 & 12 hr after first dose on Day 1; pre-dose (0 hr before morning dose) on Days 2, 3, 4, 5, 7; and pre-dose (0 hr), 0.25,0.5,1,1.5,2,3,4,6,8,10,12,24,36,48,72 & 96 hr after last morning dose on Day 14
RTV-Boosted MAD Cohort: Ctrough of RTV | Pre-dose (0 hr), 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10 & 12 hr after first dose on Day 1; pre-dose (0 hr before morning dose) on Days 2, 3, 4, 5, 7; and pre-dose (0 hr), 0.25,0.5,1,1.5,2,3,4,6,8,10,12,24,36,48,72 & 96 hr after last morning dose on Day 14
RTV-Boosted MAD Cohort: Apparent Terminal t1/2 of RTV | Pre-dose (0 hr), 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10 & 12 hr after first dose on Day 1; pre-dose (0 hr before morning dose) on Days 2, 3, 4, 5, 7; and pre-dose (0 hr), 0.25,0.5,1,1.5,2,3,4,6,8,10,12,24,36,48,72 & 96 hr after last morning dose on Day 14
RTV-Boosted MAD Cohort: Accumulation Index of RTV | Pre-dose (0 hr), 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10 & 12 hr after first dose on Day 1; pre-dose (0 hr before morning dose) on Days 2, 3, 4, 5, 7; and pre-dose (0 hr), 0.25,0.5,1,1.5,2,3,4,6,8,10,12,24,36,48,72 & 96 hr after last morning dose on Day 14

SECONDARY OUTCOMES:
MAD Cohort: Cmax of Midazolam | Pre-dose (0 hr), 0.25, 0.5,1, 2, 4, 6, 8, 10, 12, and 24 hr post-midazolam dose on Days -1 and 14
Tmax of Midazolam | Pre-dose (0 hr), 0.25, 0.5,1, 2, 4, 6, 8, 10, 12, and 24 hr post-midazolam dose on Days -1 and 14
MAD Cohort: AUC0-last of Midazolam | Pre-dose (0 hr), 0.25, 0.5,1, 2, 4, 6, 8, 10, 12, and 24 hr post-midazolam dose on Days -1 and 14
MAD Cohort: AUC0-inf of Midazolam | Pre-dose (0 hr), 0.25, 0.5,1, 2, 4, 6, 8, 10, 12, and 24 hr post-midazolam dose on Days -1 and 14
MAD Cohort: Area Under the Plasma Concentration Versus Time Curve up to 6 h Post-dose (AUC0-6h) of Midazolam | Pre-dose (0 hr), 0.25, 0.5,1, 2, 4, 6, 8, 10, 12, and 24 hr post-midazolam dose on Days -1 and 14
MAD Cohort: Apparent Terminal t1/2 of Midazolam | Pre-dose (0 hr), 0.25, 0.5,1, 2, 4, 6, 8, 10, 12, and 24 hr post-midazolam dose on Days -1 and 14
MAD Cohort: CL/F of Midazolam | Pre-dose (0 hr), 0.25, 0.5,1, 2, 4, 6, 8, 10, 12, and 24 hr post-midazolam dose on Days -1 and 14
Food-effect SAD Cohort: Cmax of RO6889678 | Pre-dose (0 hr) on Day 16; 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72 and 96 hr post Day 16 dose
Food-effect SAD Cohort: Tmax of RO6889678 | Pre-dose (0 hr) on Day 16; 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72 and 96 hr post Day 16 dose
Food-effect SAD Cohort: AUC0-last of RO6889678 | Pre-dose (0 hr) on Day 16; 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72 and 96 hr post Day 16 dose
Food-effect SAD Cohort: AUC0-inf of RO6889678 | Pre-dose (0 hr) on Day 16; 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72 and 96 hr post Day 16 dose
Food-effect SAD Cohort: Apparent Terminal t1/2 of RO6889678 | Pre-dose (0 hr) on Day 16; 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72 and 96 hr post Day 16 dose
Food-effect SAD Cohort: CL/F of RO6889678 | Pre-dose (0 hr) on Day 16; 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72 and 96 hr post Day 16 dose
Food-effect SAD Cohort: Ae of RO6889678 | Pre-dose (0 hr) on Day 16; 0-4, 4-8, 8-12, 12-24, 24-48 hours post Day 16 dose
Food-effect SAD Cohort: CLR of RO6889678 | Pre-dose (0 hr) on Day 16; 0-4, 4-8, 8-12, 12-24, 24-48 hours post Day 16 dose

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Centre For Human Drug Research; Research, Leiden, Netherlands